CLINICAL TRIAL: NCT05183763
Title: Supporting Tailored Adaptive Change and Reinforcement for Medication Adherence Program: Randomized Trial of a Novel Approach to Improve Adherence in Older Hypertensive Women and Men
Brief Title: Medication Adherence Program
Acronym: MAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Ohio State University (Other); Minds at Work (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-2221; R01HL153750 (NIH)
Record Dates: First submitted 2021-12-17; First posted 2022-01-11 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Medication Adherence; Behavior and Behavior Mechanisms
MeSH Terms: conditions — Hypertension; Medication Adherence; Behavior

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The Data Manager will calculate the primary outcome measure from pharmacy refill data prior to merging with any data file indicating group assignment. Laboratory technicians who perform the liquid chromatography tandem mass spectrometry analysis of urine metabolites of antihypertensive medications will also be blinded to group assignment. Finally, participants' primary care providers will be notified of their patients' enrollment into the study but will not be given information about group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAR-MAP (Experimental): Interactive health coaching sessions and medication reminder tools
  Interventions: Behavioral: STAR-MAP health coaching; Behavioral: Medication reminder tools
- Medication App and Reminder System Medication Adherence Program (MARS-MAP) (Active Comparator): Medication reminder tools only
  Interventions: Behavioral: Medication reminder tools

INTERVENTIONS:
Behavioral: STAR-MAP health coaching — Interactive health coaching delivered in 11 sessions over one year; focusing on using adaptive change tactics to improve medication-taking behavior
  Arms: STAR-MAP
Behavioral: Medication reminder tools — Medication-taking reminder app and pillbox

SUMMARY:
Randomized controlled trial testing the efficacy of the Supporting Tailored Adaptive change and Reinforcement for Medication Adherence Program (STAR-MAP), a health coaching approach that aims to improve antihypertensive medication adherence, blood pressure control, and quality of life. Participants (n=402) >=40 years old with a diagnosis of hypertension, uncontrolled blood pressure, and low antihypertensive medication adherence will be recruited through a statewide health insurer, Blue Cross Blue Shield of Louisiana, and randomized to receive either interactive health coaching sessions with medication reminder tools (intervention) or medication reminder tools only (control) over one year. Data will be collected from participants at baseline, 6 months, 12 months, and 24 months using questionnaires, physical measurement (height, weight, blood pressure), a computer-based single-category implicit association test, and laboratory analysis of antihypertensive medication urinary metabolites.

ELIGIBILITY:
Inclusion Criteria:

* fully insured by Blue Cross Blue Shield of Louisiana (BCBSLA)
* continuously enrolled in BCBSLA for one year
* planning to remain a member of BCBSLA for next year
* English-speaking
* telephone access
* aged ≥40 years
* diagnosis of essential hypertension (ICD-10-CM code I10)
* currently filling antihypertensive medication
* low antihypertensive medication refill (proportion of days covered (PDC) <0.8)
* low self-report adherence (4-item Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4) score ≥1)
* uncontrolled blood pressure (BP) (systolic BP ≥130 mm Hg or diastolic BP ≥80 mm Hg)
* desire to improve BP

Exclusion Criteria:

* living in a household with someone already enrolled in the study
* enrollment in another clinical trial for drug adherence or BP control
* moderate to severe cognitive impairment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion with PDC >=0.8 at 12 months | 12 months
  Proportion of days covered (PDC) calculated from pharmacy refill data

SECONDARY OUTCOMES:
Difference in mean change in PDC, baseline to 12 months | Baseline to 12 months
  Proportion of days covered (PDC) calculated from pharmacy refill data
Difference in mean change in 4-item Krousel-Wood Medication Adherence Scale score, baseline to 12 months | Baseline to 12 months
  Self-reported adherence measured by 4-item Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4; minimum value: 0 (better adherence); maximum value: 4 (worse adherence))
Difference in proportion with 4-item Krousel-Wood Medication Adherence Scale score <1 at 12 months | 12 months
  Self-reported adherence measured by 4-item Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4; minimum value: 0 (better adherence); maximum value: 4 (worse adherence))
Difference in change in proportion with high adherence as measured by urine metabolite analysis, baseline to 12 months | Baseline to 12 months
  Adherence determined by liquid chromatography tandem mass spectrometry analysis of urinary metabolites of antihypertensive medications
Difference in proportion with controlled BP at 12 months | 12 months
  Controlled blood pressure (BP) defined as systolic BP <130 mm Hg and diastolic BP <80 mm Hg; BP measured using standardized protocol
Difference in mean change in SBP, baseline to 12 months | Baseline to 12 months
  Systolic blood pressure (SBP) measured using standardized protocol
Difference in mean change in DBP, baseline to 12 months | Baseline to 12 months
  Diastolic blood pressure (DBP) measured using standardized protocol
Difference in mean change in health-related quality of life scores, baseline to 12 months | Baseline to 12 months
  Quality of life measured using 12-item Short Form Survey (SF-12); scores for eight subscales, Mental Component Summary, and Physical Component Summary calculated and compared (minimum: 0 (worse quality of life); maximum: 100 (better quality of life))

OTHER OUTCOMES:
Difference in mean change in 4-item Krousel-Wood Medication Adherence Scale score, baseline to 6 months | Baseline to 6 months
  Self-reported adherence measured by 4-item Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4; minimum value: 0 (better adherence); maximum value: 4 (worse adherence))
Difference in proportion with 4-item Krousel-Wood Medication Adherence Scale score <1 at 6 months | 6 months
  Self-reported adherence measured by 4-item Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4; minimum value: 0 (better adherence); maximum value: 4 (worse adherence))
Difference in change in proportion with high adherence as measured by urine metabolite analysis, baseline to 6 months | Baseline to 6 months
  Adherence determined by liquid chromatography tandem mass spectrometry analysis of urinary metabolites of antihypertensive medications
Difference in proportion with controlled BP at 6 months | 6 months
  Controlled blood pressure (BP) defined as systolic BP <130 mm Hg and diastolic BP <80 mm Hg; BP measured using standardized protocol
Difference in mean change in SBP, baseline to 6 months | Baseline to 6 months
  Systolic blood pressure (SBP) measured using standardized protocol
Difference in mean change in DBP, baseline to 6 months | Baseline to 6 months
  Diastolic blood pressure (DBP) measured using standardized protocol
Difference in mean change in health-related quality of life scores, baseline to 6 months | Baseline to 6 months
  Quality of life measured using 12-item Short Form Survey (SF-12); scores for eight subscales, Mental Component Summary, and Physical Component Summary calculated and compared (minimum: 0 (worse quality of life); maximum: 100 (better quality of life))
Difference in proportion with PDC >=0.8 at 24 months | 24 months
  Proportion of days covered (PDC) calculated from pharmacy refill data
Difference in mean change in PDC, baseline to 24 months | Baseline to 24 months
  Proportion of days covered (PDC) calculated from pharmacy refill data
Difference in mean change in 4-item Krousel-Wood Medication Adherence Scale score, baseline to 24 months | Baseline to 24 months
  Self-reported adherence measured by 4-item Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4; minimum value: 0 (better adherence); maximum value: 4 (worse adherence))
Difference in proportion with 4-item Krousel-Wood Medication Adherence Scale score <1 at 24 months | 24 months
  Self-reported adherence measured by 4-item Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4; minimum value: 0 (better adherence); maximum value: 4 (worse adherence))
Difference in change in proportion with high adherence as measured by urine metabolite analysis, baseline to 24 months | Baseline to 24 months
  Adherence determined by liquid chromatography tandem mass spectrometry analysis of urinary metabolites of antihypertensive medications
Difference in proportion with controlled BP at 24 months | 24 months
  Controlled blood pressure (BP) defined as systolic BP <130 mm Hg and diastolic BP <80 mm Hg; BP measured using standardized protocol
Difference in mean change in SBP, baseline to 24 months | Baseline to 24 months
  Systolic blood pressure (SBP) measured using standardized protocol
Difference in mean change in DBP, baseline to 24 months | Baseline to 24 months
  Diastolic blood pressure (DBP) measured using standardized protocol
Difference in mean change in health-related quality of life scores, baseline to 24 months | Baseline to 24 months
  Quality of life measured using 12-item Short Form Survey (SF-12); scores for eight subscales, Mental Component Summary, and Physical Component Summary calculated and compared (minimum: 0 (worse quality of life); maximum: 100 (better quality of life))

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Krousel-Wood, MD, MSPH, Principal Investigator — Tulane University
Locations (5):
- United States (5):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Tulane Doctors Dermatology & Multispecialty Clinic, Covington, Louisiana
  - Tulane Doctors Heart & Vascular and Primary Care Clinic, Metairie, Louisiana
  - Tulane University Clinical and Translational Unit, New Orleans, Louisiana
  - LSU Health Sciences Shreveport Clinical Trials Office, Shreveport, Louisiana